CLINICAL TRIAL: NCT06185309
Title: Assessment of Different Psychiatric Symptoms in Patients With Thyroid Dysfunction: Pre and Post Thyroid Treatment
Brief Title: Evaluation of Different Psychiatric Symptoms in Patients With Thyroid Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed EmadElden Mohamed, Doctor resident, Assiut University
Other Study IDs: Psychiatry & thryoid disorders
Record Dates: First submitted 2023-12-05; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Anxiety; Depression; Thyroid Dysfunction
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Evaluate psychiatric symptoms in patients with thyroid dysfunction.
2. Investigate effect of treatment on psychiatric symptoms after 2 months.

DETAILED DESCRIPTION:
Thyroid dysfunction is associated with psychiatric symptoms in addition to endocrinal manifestations.

The study aims to evaluate the prevalence of psychiatric symptoms in patients with thyroid dysfunction and investigate the response after thyroid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed as having thyroid dysfunction.

Exclusion Criteria:

* Patients with other endocrinological disorders or significant medical or neurological diseases.
* Alcohol or substance abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients newly diagnosed as having thyroid dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
The effect of thyroid treatment on psychiatric symptoms | 2 months
  Investigate the effect of thyroid treatment on psychiatric symptoms associated with thyroid dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Romany Hosny Gabra Henein, professor, Study Director — Assiut University; Khaled Ahmed Mohamed, Professor, Study Director — Assiut University

REFERENCES:
- [Result] Aslan S, Ersoy R, Kuruoglu AC, Karakoc A, Cakir N. Psychiatric symptoms and diagnoses in thyroid disorders: a cross-sectional study. Int J Psychiatry Clin Pract. 2005;9(3):187-92. doi: 10.1080/13651500510029129. PMID 24937789
- [Result] Gulseren S, Gulseren L, Hekimsoy Z, Cetinay P, Ozen C, Tokatlioglu B. Depression, anxiety, health-related quality of life, and disability in patients with overt and subclinical thyroid dysfunction. Arch Med Res. 2006 Jan;37(1):133-9. doi: 10.1016/j.arcmed.2005.05.008. PMID 16314199
- See also: Prevalence, risks, and comorbidity of thyroid dysfunction: a cross-sectional epidemiological study — https://ejim.springeropen.com/articles/10.4103/ejim.ejim_22_19